CLINICAL TRIAL: NCT06852222
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Study of Bleximenib, Venetoclax and Azacitidine for the Treatment of Participants With Newly Diagnosed Acute Myeloid Leukemia Harboring KMT2A Rearrangements or NPM1 Mutations Who Are Ineligible for Intensive Chemotherapy
Brief Title: A Study of Bleximenib, Venetoclax and Azacitidine For Treatment of Participants With Newly Diagnosed Acute Myeloid Leukemia (AML)
Acronym: cAMeLot-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 75276617AML3001; 75276617AML3001 (Other: Janssen Research & Development, LLC); 2024-520154-38-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Bleximenib and Venetoclax (VEN) + Azacitidine (AZA) (Experimental): Participants with acute myeloid leukemia (AML) will receive bleximenib in combination with venetoclax (VEN) and azacitidine (AZA) for 28-days treatment cycles and treatment will continue until progression or unacceptable toxicity.
  Interventions: Drug: Bleximenib; Drug: Venetoclax (VEN); Drug: Azacitidine (AZA)
- Arm B: Placebo and Venetoclax (VEN) + Azacitidine (AZA) (Placebo Comparator): Participants with AML will receive placebo in combination with VEN and AZA for 28-days treatment cycles, and treatment will continue until progression or unacceptable toxicity.
  Interventions: Drug: Venetoclax (VEN); Drug: Azacitidine (AZA); Drug: Placebo

INTERVENTIONS:
Drug: Bleximenib — Bleximenib will be administered orally.
  Other Names: JNJ-75276617
  Arms: Arm A: Bleximenib and Venetoclax (VEN) + Azacitidine (AZA)
Drug: Venetoclax (VEN) — VEN will be administered orally.
Drug: Azacitidine (AZA) — AZA will be administered intravenously or subcutaneously.
Drug: Placebo — Placebo will be administered orally.
  Arms: Arm B: Placebo and Venetoclax (VEN) + Azacitidine (AZA)

SUMMARY:
The purpose of this study is to assess how bleximenib and Venetoclax (VEN)+ Azacitidine (AZA) works as compared to placebo and VEN+AZA alone for the treatment of participants with newly diagnosed Acute Myeloid Leukemia (AML) with a mutation in the NPM1 or KMT2A gene.

ELIGIBILITY:
Inclusion criteria:

* Be 18 years of age or older at the time of informed consent
* Previously untreated lysine N-methyltransferase 2A gene rearranged (KMT2Ar) or nucleophosmin 1 gene mutated (NPM1m) acute myeloid leukemia (AML) with greater than or equal to (> or =) 10% bone marrow blasts per 2022 international Consensus Classification criteria
* Ineligible for intensive chemotherapy based on the following criteria: a) >= 75 years of age and ineligible per physician's discretion, with Eastern Cooperative Oncology Group (ECOG) performance status of 0-2, b) >=18 to <75 years of age with >= 1 of the following comorbidities: i) ECOG performance status of 2, ii) Severe cardiac disorder, iii) Severe pulmonary disorder, iv) Renal impairment, v) Moderate hepatic impairment vi) Comorbidity that, in the investigator's opinion, makes the participant unsuitable for intensive chemotherapy, which must be documented before enrollment as defined in the protocol. Ineligibility for intensive chemotherapy should be explicitly approved by a multidisciplinary team in countries in which this process is standard of care
* Participants must have adequate hepatic and renal function
* A female participant must agree not to be pregnant, breast-feed, plan to become pregnant and use protocol-specified contraception while enrolled in this study and for 6 months after the last dose of study treatment
* A male participant must agree to use protocol-specified contraception while enrolled in this study for at least 90 days after the last dose of study treatment
* Must sign an informed consent form indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion criteria:

* Diagnosis of acute promyelocytic leukemia (APL)
* Known active leukemic involvement of the central nervous system (CNS)
* Recipient of solid organ transplant
* Any cardiac disorders such as heart attack, uncontrolled/unstable chest pain, congestive heart failure, uncontrolled or symptomatic irregular heartbeat, blockage of a blood vessel to brain, or transient ischemic (decreased oxygen in tissue) attack within 6 months of randomization
* Active infectious hepatitis
* Live, attenuated vaccine within 4 weeks of randomization
* Known allergies, hypersensitivity, or intolerance of bleximenib, azacitidine, or venetoclax excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2029-06-22 (Estimated); Study Completion 2029-08-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Complete Remission (CR) | Up to 4 years and 1 month
  CR is defined as Bone marrow blasts less than (<) 5 percent (%); Absence of circulating blasts; Absence of extramedullary disease; Absolute neutrophil count (ANC) greater than or equal to (>=) 1.0 * 10^9/Liter (1,000/microliter [mcL]); Platelet count >= 100 * 10^9/L (100,000/mcL).
Overall Survival (OS) | Up to 4 years and 1 month
  Overall survival time is defined as the time duration from the date of randomization to death due to any cause.

SECONDARY OUTCOMES:
Event-free survival (EFS) | Up to 4 years and 1 month
  EFS is defined as the time from randomization to treatment failure, relapse, or death due to any cause, whichever occurs first.
Duration of CR | Up to 4 years and 1 month
  Duration of CR will be estimated among responders from the date of initial documentation of CR, to the date of first documented evidence of relapse, or death due to any cause, whichever occurs first, respectively.
Time to CR | Up to 4 years and 1 month
  Time to CR is defined as time from randomization to first documented response.
Rate of CR Without Measurable Residual Disease (MRD-) | Up to 4 years and 1 month
  Rate of CR MRD- is defined as percentage of participants who have achieved CR without MRD.
Percentage of Participants who Achieved Transfusion Independence | Up to 4 years and 1 month
  Transfusion independence is defined as lack of requirement for red blood cell (RBC) and platelet transfusions during any 56-day period.
Percentage of Participants with Allogeneic Hematopoietic Stem Cell Transplant (Allo-HSCT) | Up to 4 years and 1 month
  Allo-HSCT rate is defined as the percentage of participants who have undergone allo-HSCT after randomization.
Number of Participants with Adverse Events (AEs) | Up to 4 years and 1 month
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Number of Participants with Abnormalities in Clinical Laboratory Parameters | Up to 4 years and 1 month
  Participants with abnormalities in clinical laboratory parameters will be reported.
Serum Concentration of Bleximenib | Up to 4 years and 1 month
  Serum samples will be analyzed to determine concentrations of bleximenib.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (227):
- United States (38):
  - Cancer Treatment Center of America Phoenix, Goodyear, Arizona
  - University of Arkansas at Little Rock, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffit Cancer center, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - UofL Health Brown Cancer Center, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Washington University in St Louis, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - New York Presbyterian - Weill Cornell, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Einstein-Montefiore Medical Center, The Bronx, New York
  - Atrium Health, Charlotte, North Carolina
  - Novant Health, Charlotte, North Carolina
  - Novant Health, Winston-Salem, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Oncology and Hematology Care Clinic Westside, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Tennessee, Knoxville, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (6):
  - Flinders Medical Centre, Bedford Park
  - Royal Prince Alfred Hospital, Camperdown
  - St Vincents Hospital Melbourne, Fitzroy
  - St George Hospital, Kogarah
  - Peter MacCallum Cancer Centre, Melbourne
  - Princess Alexandra Hospital, Woolloongabba
- Austria (3):
  - Kepler Universitatsklinikum GmbH, Linz
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Universitaetsklinikum Salzburg Landeskrankenhaus, Salzburg
- Belgium (8):
  - AZ Sint-Jan, Bruges
  - UZ Antwerpen, Edegem
  - Ziekenhuis Oost-Limburg, Genk
  - Ghent University Hospital, Ghent
  - Chu Helora Hospital La Louviere Site Jolimont, La Louvière
  - Universitair Ziekenhuis Leuven, Leuven
  - Clinique Saint Pierre, Ottignies
  - Algemeen Ziekenhuis Delta, Roeselare
- Brazil (9):
  - Fundacao Pio XII, Barretos
  - Instituto D Or de Pesquisa e Ensino, Brasília
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Ministerio da Saude Instituto Nacional do Cancer, Rio de Janeiro
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
  - Instituto D Or de Pesquisa e Ensino, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
- Canada (8):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Cancercare Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre Victoria Hospital, London, Ontario
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
  - CIUSSS de l Est de l Ile de Montreal Installation Hopital Maisonneuve Rosemont, Montreal, Quebec
- China (25):
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The first Affiliated Hospital of Jilin University, Changchun
  - Sichuan Provincial Peoples Hospital, Chengdu
  - West China Hospital Si Chuan University, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Sun Yat Sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital Zhejiang University College of Medicine, Hangzhou
  - The First Affiliated Hospital of USTC Anhui Provincial Hospital, Hefei
  - Qilu Hospital of Shandong University, Jinan
  - The Second Hospital & Clinical Medical School Lanzhou University, Lanzhou
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Zhongda Hospital Southeast University, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Shengjing Hospital Of China Medical University, Shenyang
  - The Second People's Hospital of Shenzhen, Shenzhen
  - First Affiliated Hospital SooChow University, Suzhou
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tijian
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - TongJi Hospital of TongJi Medical College of Huazhong University of Science & Technology, Wuhan
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The first affiliated hospital of xiamen university, Xiamen
  - Henan Cancer Hospital, Zhengzhou
- Czechia (7):
  - Fakultni nemocnice Brno, Interni hematologicka a onkologicka klinika, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava - Poruba
  - Fakultni nemocnice Plzen, Pilsen
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Ustav Hematologie A Krevni Transfuze, Prague
  - Vseobecna Fakultní Nemocnice, Prague
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde
- France (12):
  - CHU d'Angers, Angers
  - CHU de Clermont Ferrand - Site Estaing, Clermont-Ferrand
  - Hopital Saint Vincent de Paul, Lille
  - Institut Paoli Calmettes, Marseille
  - CHU de Montpellier Hopital Saint Eloi, Montpellier
  - CHU De Nice Hopital De l'Archet, Nice
  - Hopital Saint Louis, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - CHU Reims Hopital Robert Debre, Reims
  - Chu Rennes Hopital Pontchaillou, Rennes
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - CHRU de Nancy - Hopitaux de Brabois, Vandœuvre Ies-Nancy
- Germany (7):
  - Klinikum Augsburg, Augsburg
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Schleswig Holstein Campus Kiel, Kiel
  - Universitaetsklinikum Leipzig, Leipzig
- Greece (7):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Evaggelismos Hospital, Athens
  - General Hospital of Athens Attikon, Chaïdári
  - University General Hospital of Ioannina, Ioannina
  - General University Hospital of Patras, Rio
  - Ahepa University General Hospital of Thessaloniki, Thessaloniki
  - Geniko Nosokomeio Thessalonikis George Papanikolaou, Thessaloniki
- Queen Mary Hospital, Hong Kong, Hong Kong
- Israel (8):
  - Shamir Medical Center Assaf Harofeh, Beer Yaakov
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospita Ein Kerem, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (13):
  - ASST Papa Giovanni XXIII Bergamo, Bergamo
  - A O U Sant Orsola Malpighi, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera di Perugia Ospedale S.Maria della Misericordia, Perugia
  - AST Pesaro e Urbino Ospedale San Salvatore, Pesaro
  - Ospedale S. Maria Delle Croci, Ravenna
  - Grande Ospedale Metropolitano 'Bianchi-Melacrino-Morelli' Reggio Calabria, Reggio Calabria
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo
- Japan (16):
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyō City
  - Kyushu University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Gifu Municipal Hospital, Gifu
  - Kanazawa University Hospital, Kanazawa
  - Kobe City Medical Center General Hospital, Kobe
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Gunmaken Saiseikai Maebashi Hospital, Maebashi
  - Nagoya University Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - Japanese Red Cross Osaka Hospital, Osaka
  - Aiiku Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Nippon Medical School Hospital, Tokyo
  - Yamagata University Hospital, Yamagata
  - University of Fukui Hospital, Yoshida
- Mexico (2):
  - Centro de Investigacion Clinica Chapultepec, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
- Poland (5):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Swietokrzyskie Centrum Onkologii SPZOZ w Kielcach, Kielce
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im M Kopernika w Lodzi, Lodz
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Portugal (5):
  - Uls Sao Jose - Hosp. Sto Antonio Dos Capuchos, Lisbon
  - Uls Santa Maria Hosp. Santa Maria, Lisbon
  - Uls Santo Antonio - Hosp. Santo Antonio, Porto
  - Instituto Portugues de Oncologia, Porto
  - Uls Sao Joao - Hosp. Sao Joao, Porto
- South Korea (7):
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (16):
  - Hosp Univ A Coruna, A Coruña
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Clinic de Barcelona, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. San Pedro de Alcantara, Cáceres
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Inst. Cat. Doncologia-H Duran I Reynals, L'Hospitalet de Llobregat
  - Clinica Univ. de Navarra, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Univ. I Politecni La Fe, Valencia
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chi Mei Medical Center Liouying Branch, Tainan
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (8):
  - Ankara Etlik Sehir Hastanesi, Ankara
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Ankara University School of Medicine Cebeci Hospital, Ankara
  - Memorial Antalya Hospital, Antalya
  - Koc University Medical Faculty, Istanbul
  - VM Medical Park Mersin Hospital, Mersin
  - Sakarya University Training and Research Hospital, Sakarya
  - Ondokuz Mayis University, Samsun
- United Kingdom (9):
  - University Hospitals Sussex NHS Foundation Trust, Brighton
  - Addenbrookes Hospital, Cambridge
  - Kent and Canterbury Hospital, Canterbury
  - Colchester Hospital University NHS, Colchester
  - Western General Hospital, Edinburgh
  - The Clatterbridge Cancer Centre, Liverpool
  - Guys' and St Thomas' NHS Trust, London
  - Derriford Hospital, Plymouth
  - University Hospitals Sussex NHS Foundation Trust, Worthing

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency